CLINICAL TRIAL: NCT05641545
Title: IVAC-RCC-001: A Personalized Neoantigen Vaccine as Add-on to Standard of Care Checkpoint Inhibitor in Advanced/Metastatic RCC Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Premature discontinuation due to üoor participant recruitment
Sponsor: SLK Kliniken Heilbronn GmbH (Other)
Responsible Party: Principal Investigator, Uwe Martens, Director of the Department of Hematology, Oncology and Palliative Care, SLK Kliniken Heilbronn GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IVAC-RCC-001
Record Dates: First submitted 2022-05-02; First posted 2022-12-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVAC-RCC-001 (Experimental): Individual peptide vaccination with adjuvant GM-CSF and Imiquimod Intradermal injection of a cocktail of 3-5 individual HLA-binding peptides. Subcutaneous injection of adjuvant GM-CSF at vaccination site. Topical administration of Imiquimod at vaccination site.
  Interventions: Biological: IVAC

INTERVENTIONS:
Biological: IVAC — IVAC is a personalized peptide vaccine

SUMMARY:
This is a monocenter, single-arm, prospective phase Ib trial, designed to evaluate the safety, clinical toxicity and in vivo immunological effects of a patient-individualized peptide vaccination added to standard of care checkpoint blockade (nivolumab) in adult patients with metastatic/advanced renal cell carcinoma who experienced at least stable disease after four cycles of standard of care immune therapy (ipilimumab/nivolumab).

DETAILED DESCRIPTION:
The aim of this clinical study is to evaluate the feasibility and safety of an individualized peptide vaccination approach in patients with advanced renal cell carcinoma who experienced at least stable disease after four cycles of standard of care immune therapy (ipilimumab/nivolumab). For this purpose, tumor-specific mutations are analyzed by comparative exome sequencing of tumor and healthy reference tissue. In a second step, HLA-binding (human leukocyte antigen-binding) peptides derived from mutated protein sequences are selected for vaccination. The peptides are administered as a vaccination cocktail with adjuvant GM-CSF and Imiquimod over a course of 9 months and a total of 16 vaccinations. Primary objective is the de novo induction of a specific T cell response without unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Ability to understand and willingness to sign a written informed consent document.
* Patients with RCC Stage IV (AJCC 8th ed.) of any histology, not amenable to curative surgery, minimal-invasive therapy or radiation therapy
* Intermediate/poor risk by IMDC (≥1 risk factors)
* ECOG 0-1
* Patients with advanced or metastatic disease occurring subsequent to initial curative nephrectomy or subsequent to other previous therapy with curative intent are eligible
* Measurable disease as per RECIST 1.1 (at least one measurable lesion)
* Participants must be eligible to be treated with first line Nivolumab+Ipilimumab based on investigator´s judgement.
* Patients must have adequate fresh tissue available. If a fresh tissue sample is not available by routine procedures, participants must have a lesion amenable to fresh tumor biopsy at study entry for the next generation sequencing (NGS) required for this study and willing to provide informed consent for such biopsy. FFPE tumor samples are not suitable for the NGS required for this study.
* Patient is agreeable to allow tumor and blood samples to be submitted for complete exome and transcriptome sequencing.
* No previous systemic therapy for advanced or metastatic RCC
* Patients with 3 or fewer brain metastases that are < 1 cm in diameter and asymptomatic are eligible if clinically stabe
* Participants must have normal organ and bone marrow function as defined below Leukocytes ≥3,000/mcL Absolute neutrophil count ≥1,000/mcL Platelets ≥100,000/mcL Total bilirubin within 1,5 ULN AST(SGOT)/ALT(SGPT) ≤5 × institutional upper limit of normal Creatinine Clearance ≥40 mL/min/(calculated using the Cockroft-Gault equation)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test before entry onto the trial and within 2 days prior to start of study medication.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity for the duration of vaccine treatment plus 30 days (duration of ovulatory cycle).

Exclusion Criteria:

* Prior treatment with any anti-programmed cell death (anti-PD-1), or anti-programmed cell death ligand 1 (anti-PD-L1) agent or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Prior systemic anti-cancer therapy for RCC with vascular endothelial growth factor (VEGF)/VEGF receptors (VEGFR) or mechanistic target of rapamycin (mTOR) targeting agents. Prior systemic anti-cancer therapy for curative intent with VEGFR or mTOR targeting agents is allowed if discontinued >6 months prior to enrolment.
* Prior RCC-directed cancer vaccine therapy.
* Any history of a known or suspected autoimmune disease [e.g. including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome) or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Participants with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Active brain metastases or leptomeningeal metastases
* Positive serological test for hepatitis C virus ot hepatitis B virus surface antigen (HBsAg) or or human immunodeficiency virus (HIV)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring IV antibiotic treatment, symptomatic congestive heart failure, unstable angina pectoris, clinically relevant cardiac arrhythmia.
* Any known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is "success of treatment" defined as a patient without unacceptable toxicity and showing a vaccination-induced T-cell response. | 120 days
  Treatment success is defined as a patient without
  1. unacceptable toxicities (grade 4 according to NCI-CTC) and in whom
  2. a vaccine-specific response of CD4+ and/or CD8+ T cells could be induced. The primary endpoint will be analyzed after 10 patients have reached visit 10

SECONDARY OUTCOMES:
To evaluate CD4+ and/or CD8+ T-cell responses over the vaccination period. | 246 days
  T-cell responses will be measured after completion of the study and will be analyzed with regard to the T-cell responses after 10 vaccinatuions /at day 120.
To evaluate the event-free survival (EFS) during and after treatment. | 246 days
  EFS will be assessed on days 120 and 246.

CONTACTS AND LOCATIONS:
Locations (1):
- SLK Kliniken Heilbronn, Klinik für Innere Medizin III: Hämatologie, Onkologie, Palliativmedizin, Heilbronn, Germany

IPD SHARING:
Plan to Share IPD: No